CLINICAL TRIAL: NCT01359969
Title: Open-label, Phase II, Single Arm Study to Evaluate the Safety, Immunogenicity, Pharmacokinetics and Efficacy of rhC1INH for the Treatment of Acute Attacks in Pediatric Patients With Hereditary Angioedema, From 2-13 Years of Age
Brief Title: Safety of Ruconest in 2-13 Year Old Hereditary Angioedema (HAE) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1 1209; 2011-000987-92 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; HAE; Angioedema; Recombinant C1 Inhibitor; rhC1INH; Pediatrics
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema | interventions — conestat alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recombinant Human C1 Inhibitor (Experimental): Patients presented to the clinic within 5 hours of onset received rhC1INH 50 U/kg body weight up to a maximum of 4200 U.
  Interventions: Drug: rhC1INH

INTERVENTIONS:
Drug: rhC1INH — Patients up to 84 kg will receive one i.v. injection of Ruconest at a dose of 50 U/kg. The reconstituted solution should be administered as a slow i.v. injection over approximately 5 minutes. Patients of 84 kg body weight or greater will receive one i.v. injection of Ruconest at the dose of 4200 U (2 vials).
  Other Names: Ruconest

SUMMARY:
This open-label study is being conducted to confirm the safety, pharmacokinetic profile and efficacy of Ruconest at a dose of 50 U/kg when used for the treatment of acute angioedema attacks in patients, from 2 up to and including 13 years of age.

DETAILED DESCRIPTION:
This study was an open-label, Phase 2, non-comparative, multinational, multicenter clinical study in pediatric patients from 2 up to and including 13 years of age, with a confirmed diagnosis of HAE. Patients were eligible for treatment with recombinant human C1-inhibitor (rhC1INH) if they presented to the clinic within 5 hours of onset with an acute attack of at least moderate severity without signs of spontaneous regression. Patients received rhC1INH at a dose of 50 U/kg body weight up to a maximum of 4200 U. The reconstituted solution was administered as a slow intravenous (iv) injection over approximately 5 minutes. The patients remained in hospital and were closely monitored in the study center for at least 4 hours after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* From 2 up to and including 13 years of age
* Clinical and laboratory confirmed diagnosis of HAE (baseline C1INH activity <50% of normal)
* Signed written Informed Consent Form (ICF)(parental permission) signed by the legal guardian(s)
* Clinical symptoms of an acute HAE attack
* Onset of eligible symptoms within 5 hours from the moment at which medical evaluation to determine eligibility has occurred
* Attack severity moderate or greater, as rated by the investigator

Exclusion Criteria:

* A diagnosis of acquired C1INH deficiency (AAE)
* A medical history of allergy to rabbits or rabbit-derived products or positive anti-rabbit epithelium (dander) immunoglobuline E (IgE) test

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Relan, MD, Study Director — VP Clinical Research & Medical Affairs at Pharming
Locations (16):
- Portland Clinical Research/AAIM Care, LLC, Portland, Oregon, United States
- Czechia (2):
  - UIA FN Plzen ( Institute of Immunology and Allergology), Faculty Hospital Plzen, Pilsen, Alej Svobody 80
  - University Hospital Motol, Institute of Immunology, Prague, V Úvalu 84
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin, Charitéplatz 1
  - Klinikum Rechts der Isar, Technical University Munich, Munich
- Heim Pál Gyermekkórház, II. számú Gyermek Belgyógyászati Osztály, Budapest, Madarász Utca 22-24, Hungary
- Israel (3):
  - Bnei Zion Hospital, Haifa
  - Souraski Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (2):
  - Hospital Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria S. Giovanni di Dio e Ruggi d'Aragona, Salerno
- University Clinic Of Dermatology Skopje, Skopje, North Macedonia
- Poland (2):
  - Pediatric Hospital, Krakow
  - Pediatric Hospital, Lublin
- Mures County Clinical Hospital, Târgu Mureş, Romania
- Klinika detí a dorastu, Univerzitna nemocnica Martin, Martin, Kollárova 2, Slovakia

REFERENCES:
- [Result] Reshef A, Grivcheva-Panovska V, Kessel A, Kivity S, Klimaszewska-Rembiasz M, Moldovan D, Farkas H, Gutova V, Fritz S, Relan A, Giannetti B, Magerl M. Recombinant human C1 esterase inhibitor treatment for hereditary angioedema attacks in children. Pediatr Allergy Immunol. 2019 Aug;30(5):562-568. doi: 10.1111/pai.13065. Epub 2019 May 29. PMID 30993784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female patients, from 2 up to and including 13 years of age with a clinically suspected and/or confirmed diagnosis of HAE will be recruited for this study. Patients will be identified and invited to participate by the investigators at the respective study centers.
Pre-assignment Details: Screening details:
  Pts with a med hist of HAE (age 2-13 yrs) were invited for a screening visit. At screening the diagnosis HAE was confirmed via Central lab testing. If the diagnosis was confirmed, pts were eligible for treatment if an acute attack would occur and they presented to study center within 5 hrs of onset of attack. In total 57 pts signed ICF and 20 pts had one or more HAE attacks treated.
Period: Overall Study
Arm/Group | Recombinant Human C1 Inhibitor
Started | 57 (The study continued until at least 20 patients had been treated with rhC1INH for at least one acute HAE attack. 57 patients were eligible for treatment and included in the Screening Analysis Set, 37 enrolled patients had no attack and therefore no treatment.)
Completed | 20
Not Completed | 37
Not completed — Study continued until at least 20 patients had been treated for at least one treatment. | 37

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 9.55 (3.304)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Romania | 2
  Hungary | 1
  Czechia | 2
  United States | 1
  Poland | 2
  North Macedonia | 2
  Israel | 9
  Germany | 1
Height at screening [Mean (Standard Deviation); unit: centimeters] | 125.6 (25.78)
Weight at presentation [Mean (Standard Deviation); unit: kilograms] | 34.81 (20.554)

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Relief Based on Visual Analogue Scale (VAS) Was Defined as the Time, in Minutes, From Time of Infusion to the Beginning of Relief.
Description: Time to beginning of relief of symptoms that showed the response to treatment based on the overall VAS score decrease of ≥ 20 mm from baseline. Separate VAS forms will be given to express the current feelings considering the severity of angioedema symptoms for five possible anatomical locations. The form will be completed by placing vertical marks on each of the 100 mm horizontal lines. The Abdominal VAS measures the patient's perceptions relating to illness, pain, bloodedness, and nausea; the oro-pharyngeal-laryngeal (OPL) VAS measures illness, pain, swelling, breathing, speech, and swallowing; the facial VAS instrument measure illness, pain and swelling; the Peripheral VAS measures swelling, pain, and use of extremity; and the Urogenital VAS measures illness, pain, swelling, nausea, and urination. Time to beginning of relief will also be calculated based on the Investigator Score (IS) and Treatment Effect Questionnaire (TEQ).
Time Frame: The assessment of the angioedema signs by the VAS and TEQ will be performed just before start of infusion, and at T30m, T1h, T2h, T4h, T8h and T24h after study medication infusion VAS score decrease of ≥ 20 mm from baseline.
Population: No statistical analyses have been specified for this primary end point. As this was an open-label single arm study, no statistical analyses could be provided.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 20
minutes | 60 [60 to 65]

2. Secondary Outcome: Time to Minimal Symptoms Based on Patient's VAS Scores; Time From the Start of the Infusion of Study Medication to the First Assessment Time at Which the Overall Severity VAS Reaches a Value of Less Than 20 mm for All Locations
Description: Time to minimal symptoms was defined as the time at which the Overall VAS score fell below 20 mm for all locations where VAS Scores were recorded. Separate VAS forms will be given to express the current feelings considering the severity of angioedema symptoms for five possible anatomical locations. The form will be completed by placing vertical marks on each of the 100 mm horizontal lines provided to answer each question related to the severity of symptoms and the patient's condition. The Abdominal VAS measures the patient's perceptions relating to illness, pain, bloodedness, and nausea; the OPL VAS measures illness, pain, swelling, breathing, speech, and swallowing; the facial VAS instrument measure illness, pain and swelling; the Peripheral VAS measures swelling, pain, and use of extremity; and the Urogenital VAS measures illness, pain, swelling, nausea, and urination.
Time Frame: The assessment of the angioedema signs by the VAS and TEQ will be performed just before start of infusion, and at T30m, T1h, T2h, T4h, T8h and T24h after study medication infusion all locations where VAS Scores were recorded.
Population: No statistical analyses for this end point
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Recombinant Human C1 Inhibitor
Number analyzed (Participants) | 20
minutes | 122.5 [120 to 126]

ADVERSE EVENTS:
Time Frame: Investigators are required to document all AEs occurring during the clinical study, commencing with the signing of the ICF through the last follow-up visit (Day 90 after the last treatment).
Description: The reported values are based on the treatment-emergent (serious) adverse events (TE(S)AE), which are the (S)AEs with an onset at any time between the start of treatment and 97 days after treatment for any treated attack. The AEs are only analyzed for the 20 treated patients. The TLFs are based on these 20 treated and analyzed patients. A total of 11 patients experienced 30 TEAEs after treatment with rhC1INH. A total of 3 patients experienced 9 TESAEs after treatment with rhC1INH.
Arm/Group | Recombinant Human C1 Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human C1 Inhibitor (N=20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human C1 Inhibitor (N=20)
Lymphocyte morphology abnormal (Vascular disorders) | 2 (2)
Pallor (Vascular disorders) | 1 (1)
Body temperature increased (Vascular disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT01359969/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT01359969/SAP_001.pdf